CLINICAL TRIAL: NCT02715232
Title: Effects of Sex Steroid Hormones on Serotonin Synthesis and Degradation Measured With PET
Brief Title: Effects of Sex Steroids on the Serotonin System
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc. Prof., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1.1-20150511
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria | interventions — Testosterone; Lynestrenol; Cyproterone Acetate; Estradiol; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female-to-Males (Experimental): Female-to-Male Transsexuals receiving Testosterone treatment
  Interventions: Drug: Testosterone; Drug: Lynestrenol; Drug: Triptorelin acetate
- Male-to-Females (Experimental): Male-to-Female Transsexuals receiving Estradiol and Anti-androgen treatment
  Interventions: Drug: Cyproterone Acetate; Drug: Estradiol; Drug: Triptorelin acetate
- Female Controls (No Intervention): Female Controls receiving no intervention
- Male Controls (No Intervention): Male controls receiving no intervention

INTERVENTIONS:
Drug: Testosterone — 100mg testosterone undecanoat every 8-12 weeks, or alternatively 50mg testosterone transdermally, or 50mg testosterone creme
  Arms: Female-to-Males
Drug: Lynestrenol — 2-3 tablets/day, if menstruation still occurs
  Arms: Female-to-Males
Drug: Cyproterone Acetate — 25mg daily
  Arms: Male-to-Females
Drug: Estradiol — 75 microgram transdermal therapeutic system twice a week, or p.o. estradiol 2x2mg/day, or estradiol gel 1,5-3mg
  Arms: Male-to-Females
Drug: Triptorelin acetate — 4,12mg every 4-6 weeks (powder for suspension for injection s.c. or i.m.
  Arms: Female-to-Males; Male-to-Females

SUMMARY:
The aim of this study is to prove the modulatory influence of sex hormones on serotonergic neurotransmission by determining the enzymatic processes involved in serotonin synthesis and degradation using positron emission tomography (PET) in humans in vivo with the radiotracers [11C]AMT and [11C]harmine.

DETAILED DESCRIPTION:
Background:

Sex hormones such as estradiol and testosterone modulate human brain structure and function and are tightly connected to neuropsychiatric disorders such as depression and anxiety disorders. Using molecular imaging in humans in vivo, the investigators showed strong influences of sex hormones on serotonergic neurotransmission via modulation of serotonergic receptors and transporters. Although, animal studies also indicate strong modulatory influences on serotonin synthesis and degradation, human data on this potential effect are absent.

Objectives of the study:

The aim of this study is to prove the modulatory influence of sex hormones on serotonergic neurotransmission by determining the enzymatic processes involved in serotonin synthesis and degradation using positron emission tomography (PET) in humans in vivo with the radiotracers [11C]AMT and [11C]harmine.

Study design:

Single-blind, longitudinal study. Transsexuals will undergo four PET and two magnetic resonance imaging (MRI) measurements: 1. One [11C]AMT PET, one [11C]harmine PET and one MRI measurement before start of treatment, 2. One [11C]AMT PET, one [11C]harmine PET and one MRI measurement after 4 months of treatment. The investigators propose an overall study duration of 36 months.

Materials and Methods:

PET measurements will be performed on a GE Advance PET scanner. To examine the interdependence between serotonin activity and brain structure and function, four MRI sequences will be performed in order to assess gray matter volume and cortical thickness, gray and white matter microstructure, as well as resting state functional connectivity and cerebral blood flow. MRI measurements will be done on a 3 Tesla scanner with high spatial and temporal resolution.

Study population:

20 healthy female-to-male (FtM), 20 healthy male-to-female (MtF) transsexuals (aged 18-50) who are free of hormone-medication at baseline; 40 healthy controls, matched for sex, age and education level.

Pilot Study:

A pilot study without pharmacologic intervention consisting of one optional [11C]AMT PET and two [11C]harmine PET will be performed in 12 healthy controls in order to optimise PET measurement procedures.

Relevance and implications of the study:

This will be the first imaging study to investigate the effects of high-dose, long-term opposite-sex steroid hormones on serotonin synthesis and degradation in the living human brain using PET. The study will lead to the establishment of a comprehensive theory of serotonergic modulation by sex steroids and will increase knowledge on the serotonergic role in shaping brain morphology, microstructure and structural/functional connectivity. Results will provide essential data for a better understanding of neural sex differences associated with differences in hormonal states in humans and will elucidate neurobiological correlates of the known gender difference in the prevalence of neuropsychiatric disorders, thus contributing to the development of personalized treatment, the reduction of personal suffering and the reduction of costs and occupational disability.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of Gender Dysphoria (DSM-5: 302.85; ICD-10: F64.1) (for transsexuals only)
* Somatic health based on history, physical examination, ECG, laboratory screening, SCID
* willingness and competence to sign the informed consent form

Exclusion Criteria:

* concomitant major medical or neurological illness
* internal or neurologic medical histories as well as pregnancy (positive urine pregnancy test) or breastfeeding
* other DSM-5 Axis-I comorbidities, determined by a structured clinical interview (SCID), especially body dysphoric disorder (DSM-5: 300.7; ICD-10: F45.22), schizophrenia spectrum and other psychotic disorders
* steroid hormone treatment within 6 months prior to inclusion
* treatment with psychotropic agents such as SSRIs
* any implant or stainless steel graft
* abnormal values in routine laboratory screening or general physical examination
* current substance abuse or current or past substance related disorder
* for participants who participated in an earlier neuroimaging study using ionizing radiation, the total radiation exposure dose of 20 mSv over the last 10 years must not be exceeded, as specified in the legislation on radiation protection (Allg. Strahlenschutzverordnung 2010; www.ris.bka.gv.at)
* failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
blood-to-brain clearance/trapping (K*) of [11C]AMT | <5 months
  [11C]AMT trapping as an estimation of brain serotonin synthesis in vivo in humans
distribution volume (DV) of [11C]harmine | <5 months
  distribution volume of specifically bound radioligand [11C]harmine in brain regions

SECONDARY OUTCOMES:
white and gray matter microstructure | <5 months
  microstructure measured using diffusion weighted imaging
gray matter volume/density and cortical thickness | <5 months
  structural MRI measurements
cerebral blood flow (CBF) | <5 months
  cerebral blood flow measured using arterial spin labeling MRI
Scores on the Klein Sexual Orientation Grid (KSOG) | <5 months
  the KSOG measures sexual orientation
Scores on the Utrecht Gender Dysphoria Scale | <5 months
  Score for gender dysphoria

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, MD, Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kranz GS, Wadsak W, Kaufmann U, Savli M, Baldinger P, Gryglewski G, Haeusler D, Spies M, Mitterhauser M, Kasper S, Lanzenberger R. High-Dose Testosterone Treatment Increases Serotonin Transporter Binding in Transgender People. Biol Psychiatry. 2015 Oct 15;78(8):525-33. doi: 10.1016/j.biopsych.2014.09.010. Epub 2014 Sep 23. PMID 25497691
- [Background] Kranz GS, Hahn A, Kaufmann U, Kublbock M, Hummer A, Ganger S, Seiger R, Winkler D, Swaab DF, Windischberger C, Kasper S, Lanzenberger R. White matter microstructure in transsexuals and controls investigated by diffusion tensor imaging. J Neurosci. 2014 Nov 12;34(46):15466-75. doi: 10.1523/JNEUROSCI.2488-14.2014. PMID 25392513
- [Background] Hahn A, Kranz GS, Kublbock M, Kaufmann U, Ganger S, Hummer A, Seiger R, Spies M, Winkler D, Kasper S, Windischberger C, Swaab DF, Lanzenberger R. Structural Connectivity Networks of Transgender People. Cereb Cortex. 2015 Oct;25(10):3527-34. doi: 10.1093/cercor/bhu194. Epub 2014 Sep 12. PMID 25217469
- [Background] Hahn A, Kranz GS, Sladky R, Kaufmann U, Ganger S, Hummer A, Seiger R, Spies M, Vanicek T, Winkler D, Kasper S, Windischberger C, Swaab DF, Lanzenberger R. Testosterone affects language areas of the adult human brain. Hum Brain Mapp. 2016 May;37(5):1738-48. doi: 10.1002/hbm.23133. Epub 2016 Feb 15. PMID 26876303
- [Background] Smith LJ, Henderson JA, Abell CW, Bethea CL. Effects of ovarian steroids and raloxifene on proteins that synthesize, transport, and degrade serotonin in the raphe region of macaques. Neuropsychopharmacology. 2004 Nov;29(11):2035-45. doi: 10.1038/sj.npp.1300510. PMID 15199371
- [Background] Aggarwal M, Puri V, Puri S. Effects of estrogen on the serotonergic system and calcitonin gene-related peptide in trigeminal ganglia of rats. Ann Neurosci. 2012 Oct;19(4):151-7. doi: 10.5214/ans.0972.7531.190403. PMID 25205989
- [Background] Purves-Tyson TD, Handelsman DJ, Double KL, Owens SJ, Bustamante S, Weickert CS. Testosterone regulation of sex steroid-related mRNAs and dopamine-related mRNAs in adolescent male rat substantia nigra. BMC Neurosci. 2012 Aug 6;13:95. doi: 10.1186/1471-2202-13-95. PMID 22867132
- [Derived] Klobl M, Reed MB, Handschuh P, Kaufmann U, Konadu ME, Ritter V, Spurny-Dworak B, Kranz GS, Lanzenberger R, Spies M. Gender Dysphoria and Sexual Euphoria: A Bayesian Perspective on the Influence of Gender-Affirming Hormone Therapy on Sexual Arousal. Arch Sex Behav. 2024 May;53(5):1859-1871. doi: 10.1007/s10508-023-02778-1. Epub 2024 Jan 12. PMID 38216784